CLINICAL TRIAL: NCT02290457
Title: Effects of Core Strength Training Using Unstable Surfaces on Physical Fitness in Adolescents
Brief Title: Core Strength Training in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Potsdam (Other)
Collaborators: THIM - die internationale Hochschule für Physiotherapie (Other); Free University of Brussels (Other)
Responsible Party: Principal Investigator, Urs Granacher, Prof. Dr., University of Potsdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPotsdam
Record Dates: First submitted 2014-11-10; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Exercise; Strength Training
Keywords: resistance training; trunk muscle strength; physical fitness; adolescent
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSTS (Experimental): core strength training performed on stable surfaces
  Interventions: Behavioral: core strength training
- CSTU (Experimental): core strength training performed on unstable surfaces
  Interventions: Behavioral: core strength training

INTERVENTIONS:
Behavioral: core strength training — Both training programs will last 6 weeks and comprise 2 training sessions per week with a total of 12 training sessions for each intervention group. Each training session will last 30 min, starting with a brief warm-up program mainly consisting of core strength exercises at moderate intensities and ending with a cool-down program (i.e., dynamic stretching). During the main part of training, both groups mainly conduct the "big 3" exercises as described by McGill. These will include the curl-up, side bridge, and quadruped position. In other words, every single training session will consist of frontal, dorsal, and lateral core exercises. The only difference between the 2 intervention groups is that the CSTU protocol comprise core exercises that will be conducted on unstable elements (e.g., TOGU© DYNAIR PRO, THERA-BAND© STABILITY TRAINER), whereas the CSTS program will contain the same exercises on stable surface only.

SUMMARY:
Background: It has been demonstrated that core strength training is an effective means to enhance trunk muscle strength (TMS) and athletic performance in youth. However, the role of instability with core strength training is unresolved in youth. This study specifically will investigate the effects of core stability (CST) compared to core instability strength training (CIST) on physical fitness in adolescents.

Methods: Twenty-seven (14 girls, 13 boys) healthy adolescents (age 14±1 years) will be assigned to a CST (n=13) or a CIST (n=14) group. Both training programs will last 6 weeks (2 sessions/week) and included frontal, dorsal, and lateral core exercises. During CIST, these exercises will be conducted on unstable surfaces (e.g., TOGU© DYNAIR CUSSIONS, THERA-BAND© STABILITY TRAINER).

Expected Results: Based on selected results reported in the literature, we hypothesize that participants performing CIST as compared to CST will show larger improvements in physical fitness tests (i.e., strength, speed, flexibility, coordination, balance) following training. Of note, training induced gains in strength, speed, flexibility, coordination, and balance are of vital importance for sports performance, everyday activities, and injury prevention.

DETAILED DESCRIPTION:
Adaptations following core strength training performed on stable (CST) as compared to unstable surface conditions (CIST) will be assessed in a pre- versus post-test design. The training period will last 6 weeks to induce training induced changes in measures of strength, speed, flexibility, coordination, and balance. These health (i.e., strength, flexibility) and skill-related (i.e., balance, coordination, speed) components of physical fitness will be assessed using physical fitness tests (i.e., Bourban TMS test, standing long jump test, 20-m sprint test, stand-and-reach test, jumping sideways test, Emery balance test, Y balance test).

Twenty-seven healthy adolescent boys and girls will participate in this study after the experimental procedures were explained. An a priori power analysis with an assumed Type I error of 0.05 and a Type II error rate of 0.20 (80% statistical power) was calculated for measures of trunk muscle strength and revealed that 13 participants per group would be 105 sufficient to observe medium Test x Group interaction effects. Study participants will be recruited from local sports clubs.

Both core strength training programs will be supervised and conducted by 2 experienced physiotherapists. The two programs will be organized as circuit training with each instructor supervising 6-7 participants. Both training programs will comprise 2 training sessions per week with a total of 12 training sessions for each intervention group. Each training session will last 30 min, starting with a brief warm-up program mainly consisting of core strength exercises at moderate intensities and ending with a cool-down program (i.e., dynamic stretching). During the main part of training, both groups mainly conduct the "big 3" exercises as described by McGill. These include the curl-up, side bridge, and quadruped position. In other words, every single training session will consist of frontal, dorsal, and lateral core exercises. The only difference between the 2 intervention groups is that the CIST protocol comprised core exercises that will be conducted on unstable elements (e.g., TOGU© DYNAIR PRO, SENSO, TOGU© REDONDO BALLS, TOGU© POWERBALLS, THERA-BAND© STABILITY TRAINER, THERA-BAND© EXERCISE BALL), whereas the CST program will contain the same exercises on stable surface only.

Prior to testing, all participants will perform a standardized 5-minutes warm-up which consists of bipedal and monopedal balance, submaximal plyometric, and skipping exercises. Thereafter, physical fitness tests (i.e., Emery balance test, Y balance test, stand-and-reach test, 20-m sprint test, jumping sideways test, standing long jump test, Bourban TMS test) will be assessed.

A multivariate analysis of variance (MANOVA) will be used to detect differences between study groups in all baseline variables. The effects of core strength training on variables of physical fitness will be analysed in separate 2 (Group: CST, CIST) x 2 (Test: pre, post) ANOVA with repeated measures on test. When Test x Group interactions reached the level of significance, group-specific post hoc tests (i.e., paired t-tests) will be conducted to identify the comparisons that were statistically significant. Additionally, the classification of effect sizes (f) will be determined by calculating partial eta squared.

ELIGIBILITY:
Inclusion Criteria:

* healthy; physically active

Exclusion Criteria:

* musculoskeletal, neurological or orthopaedic disorders that might affect their ability to perform physical fitness tests and core strength training

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Bourban trunk muscle strength (TMS) test | approx. 20 min.
  The Bourban TMS test assesses core strength endurance of ventral, lateral, and dorsal trunk muscle chains.

SECONDARY OUTCOMES:
Standing long jump test | approx. 5 min.
  Subjects will e instructed to stand with both feet right behind a starting line and to jump as far as possible. Subjects will be allowed to use arm swing during the test.
20-m sprint test | approx. 5 min.
  Subjects will be instructed to stand with one foot right behind the starting line and to accelerate at maximum effort to the finish line.
stand-and-reach test | approx. 3 min.
  Subjects will be instructed to begin the test in a standing position on an elevated platform with feet together. They will be asked to bend over using their maximal range of motion. During the test, knees, arms, and fingers will be fully extended.
jumping sideways test | approx. 5 min.
  Subjects will be instructed to jump as many times as possible over a period of 15 s with both legs together back and forth across a strip of wood that was attached to a mat (50 x 100 cm). The number of jumps completed without touching the strip and without stepping off the mat will be used as dependent variable.
Emery balance test | approx. 10 min.
  The Emery balance test will be conducted barefooted in single leg stance on an Airex balance pad. Eyes will be closed and both legs will be tested. For experimental testing, participants will be asked to stand as stable as possible with the knee of the weight-bearing limb flexed at 30°. The non-weight-bearing limb will be flexed 45° at the knee and hands will be placed on hips. Using a stopwatch, time will be stopped upon loss of balance to the nearest 1/100 of a second and will be used as dependent variable.
Y balance test | approx. 20 min.
  The lower quarter Y balance test is a dynamic test that requires subjects to maintain single leg stance while reaching as far as possible with the contralateral leg in 3 different movement directions (i.e., anterior, posteromedial, posterolateral). Subjects will always start with the right foot placed at the centre of the grid and the left leg reaching in anterior direction as far as possible, lightly touching the farthest point possible on the line with the most distal part of the reach foot. Participants will then return to a bilateral stable stance position. After 3 reaches, the left foot will be placed at the centre of the grid and the right leg will be maximally reached in anterior direction. Thereafter, the same test procedure will be conducted for the posteromedial and the posterolateral reach.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Granacher, PhD, Principal Investigator — University of Potsdam

REFERENCES:
- [Derived] Granacher U, Schellbach J, Klein K, Prieske O, Baeyens JP, Muehlbauer T. Effects of core strength training using stable versus unstable surfaces on physical fitness in adolescents: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2014 Dec 15;6(1):40. doi: 10.1186/2052-1847-6-40. eCollection 2014. PMID 25584193